CLINICAL TRIAL: NCT05197023
Title: A RANDOMIZED, DOUBLE-BLIND, DOSE-ESCALATION, PLACEBO-CONTROLLED PHASE I CLINICAL STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF MULTIPLE SUBCUTANEOUS INJECTIONS OF SHR-1819 IN PATIENTS WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: A STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF MULTIPLE SUBCUTANEOUS INJECTIONS OF SHR-1819 IN PATIENTS WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR-1819-103
Record Dates: First submitted 2021-11-26; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-11

CONDITIONS: Moderate to Severe Atopic Dermatitis

STUDY DESIGN:
Intervention Model Description: SHR1819 injection dose-escalation in AD patients
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1819 injection (Experimental)
  Interventions: Drug: SHR-1819 injection or placebo
- placebo (Placebo Comparator)
  Interventions: Drug: SHR-1819 injection or placebo

INTERVENTIONS:
Drug: SHR-1819 injection or placebo — Drug: SHR-1819 injection or placebo Low-dose group, once per week Drug: SHR-1819 injection or placebo High-dose group, once per week

SUMMARY:
The study will be conducted to evaluate the safety and tolerability of SHR-1819 injection and describe the PK/PD/ADA and explore the clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form prior to starting any study-related procedures, be able to communicate with the investigator, understand and be willing to complete this study in strict accordance with the requirements of the study protocol;
2. Age ≥ 18 years and ≤ 65 years on the day of signing informed consent form, male or female;
3. Have been diagnosed with atopic dermatitis (as per American Academy of Dermatology Criteria[6], 2014) for at least 1 year prior to screening;
4. Have moderate to severe atopic dermatitis during screening and baseline periods. Moderate to severe disease is defined as meeting the following 3 conditions at the same time:

1) Eczema Area and Severity Index (EASI) score ≥ 12; 2) Investigator's Global Assessment (IGA) score ≥ 3; 3) Body Surface Area Involvement of Atopic Dermatitis (BSA) ≥ 10%; 5. Subjects must meet at least one of the following conditions within 6 months prior to screening, as judged by the investigator:

1. Inadequate response to stable treatment with topical corticosteroids (TCS) and/or topical calcineurin inhibitors (TCI) for at least 4 weeks;
2. Or inadequate response to longest duration of treatment recommended by the prescribing information of a topical medication (such as: 14 days of treatment with super potent TCS);
3. Or unsuitable for topical treatment as judged by the investigator (such as intolerable or with contraindications); 6. Have used stable doses of basic, mild, topical emollient (moisturizer) without active ingredients twice daily for at least 7 consecutive days prior to baseline period, and continue to use during the study; 7. Subjects (including their partners) must have no fertility plan and agree to adopt effective contraceptive measures throughout the study (starting from 2 weeks before the first dose for female subjects) until 4 months after the last dose. Male subjects must agree to use a condom during intercourse throughout the study until 4 months after the last dose; female subjects of childbearing potential must have a negative human chorionic gonadotropin (HCG) test result during screening or baseline period, not be breastfeeding, and only be enrolled after confirmation of the last menstruation; female subjects without childbearing potential, the definition of without childbearing potential is: permanent sterilization (such as bilateral oophorectomy, hysterectomy, bilateral salpingectomy) or menopausal women (defined as more than 12 months of amenorrhea without pathological etiology and serum follicle-stimulating hormone (FSH) > 40 IU/L).

Exclusion Criteria:

-

General conditions:

1. Pregnant or lactating women (pregnancy is defined as the state from conception to termination of gestation) or tested positive for human chorionic gonadotropin (HCG);
2. Have a history of alcohol abuse or illegal drug abuse within 6 months prior to screening;
3. Have conditions that may affect the safety and efficacy evaluations of the investigational product based on the investigator's judgment; 2. Laboratory test results and/or 12-lead ECG findings during the screening or baseline period (tests may be repeated one time for confirmation when necessary):

1) Hemoglobin < 100.0 g/L (male) or < 90.0 g/L (female); 2) White blood cell count < 3.0 × 109/L; 3) Neutrophil count < 1.5 × 109/L; 4) Platelet count < 100 × 109/L; 5) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN); 6) Total bilirubin (T-BIL) > 1.5 × ULN; 7) Serum creatinine > ULN; 8) Positive for hepatitis B surface antigen (HBsAg), human immunodeficiency virus antibody (HIV), syphilis antibody, or hepatitis C virus (HCV) antibody; 9) Clinically significant abnormal 12-lead ECG findings that may affect the subject safety, including but not limited to acute myocardial ischemia, myocardial infarction, severe arrhythmia, or significant QTc prolongation (QTc > 500 ms).

3. Have any of the following medical histories or concurrent diseases:

1. Allergy to investigational product or any component of the investigational product;
2. History of vernal keratoconjunctivitis (VKC) and/or atopic keratoconjunctivitis (AKC);
3. Known or suspected history of immunosuppression, including a history of invasive opportunistic infections (such as tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis), even if the infection has resolved; or abnormally frequent, recurrent, or long-term infection based on the investigator's judgment;
4. active chronic active or acute infection requiring systemic treatments such as antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to screening; or superficial skin infection within 1 week prior to screening. Note: A patient may be re-screened (once only) after the infection has resolved;
5. Diagnosed with or suspected of active tuberculosis, latent untreated tuberculosis, incompletely treated tuberculosis, or nontuberculous mycobacterial infection based on the investigator and/or infectious disease specialist's judgment (as indicated by medical history, symptoms, signs, laboratory tests, X-ray or CT findings) (except subjects with treatment records demonstrating adequate treatment, who may begin treatment with biological product based on the investigator and/or infectious disease specialist's judgment);
6. History of parasite infestation/infection within 6 months prior to screening;
7. Prior (within 5 years prior to screening) or current malignant tumors (except for completely resected squamous cell carcinoma of skin, basal cell carcinoma, or cervical carcinoma in situ with no evidence of recurrence);
8. Severe, progressive, and uncontrolled cardiovascular, cerebrovascular, hepatic, renal, lung, gastrointestinal, hematopoietic, endocrine, nervous system, and psychiatric disorders, as well as other conditions that are unsuitable for study participation, as judged by the investigator.

4. Used any of the following drugs/treatments or participated in a clinical study (defined as having signed informed consent form and received treatment with a drug/medical device at least once): Received treatment with other biological products targeting IL-4Rα or participated in a clinical study involving another biological product targeting IL-4Rα;

1. Received treatment with an investigational drug (such as JAK inhibitors) or medical device within 8 weeks or 5 half-lives prior to baseline (whichever is longer);
2. Received treatment with systemic corticosteroids or immunosuppressants for atopic dermatitis within 4 weeks prior to baseline;
3. Received systemic treatment with Traditional Chinese medicine for atopic dermatitis within 4 weeks prior to baseline;
4. Received ultraviolet phototherapy (including but not limited to narrow-band ultraviolet B phototherapy (NB-UVB) and medium- to high-dose UVA1) or regular use of tanning booth/parlor for atopic dermatitis within 4 weeks prior to baseline;
5. Used bleach baths ≥ 2 times within 2 weeks prior to baseline;
6. Received the following topical medications for atopic dermatitis within 1 week prior to baseline:

   1. Topical corticosteroids or topical calcineurin inhibitors;
   2. Topical traditional Chinese medicine;
   3. Other topical medications (including but not limited to phosphodiesterase 4 (PDE-4) inhibitor);
7. Received treatment with the following biological products prior to baseline:

   1. Any cell depletion therapy, including but not limited to rituximab: within 6 months prior to baseline or until lymphocyte count returns to normal (whichever is longer);
   2. Other biological products: within 5 half-lives (if the half-life is known) or 16 weeks prior to baseline (whichever is longer);
8. Received allergen-specific immunotherapy within 6 weeks prior to baseline;
9. Received treatment with leukotriene inhibitors within 4 weeks prior to baseline;
10. Started treatment with prescription emollients or emollients containing active ingredients (such as ceramide, hyaluronic acid, urea, or filaggrin breakdown products) during the screening period (patients may continue to use these types of emollients at stable doses if they have already been using them prior to the screening visit);
11. Underwent major surgery within 3 months prior to baseline or have not recovered, or plan to undergo major surgery during the course of the study;
12. History of blood donation or severe blood loss (total blood loss ≥ 500 mL) within 1 month prior to screening, or received blood transfusion within 2 months prior to screening;
13. Received a live attenuated vaccine/live vaccine within 12 weeks prior to baseline, or plan to receive a live attenuated vaccine/live vaccine during the course of the study, or participated in a vaccine clinical trial within 12 weeks prior to baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06-08 (Estimated); Study Completion 2022-06-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) | Baseline up to end of study (up to Day 85)

SECONDARY OUTCOMES:
Pharmacokinetics of Dupilumab: Peak Plasma Concentration (Cmax) | 1-85 days
Pharmacokinetics of Dupilumab: Area under the plasma concentration versus time curve(AUC) | 1-85 days
Pharmacokinetics of Dupilumab: Elimination half life (t1/2) | 1-85 days
Pharmacokinetics of Dupilumab: Apparent clearance(CL/F) | 1-85 days
Pharmacokinetics of Dupilumab: Apparent volume of distributions(VZ/F) | 1-85 days
Pharmacokinetics of Dupilumab: Trough concentration(Ctrough) | 1-85 days
Serum TARC level and its percentage change from baseline | 1-85 days
Serum CCL17 level and its percentage change from baseline | 1-85 days
Serum immunoglobulin E (IgE) level and its percentage change from baseline | 1-85 days
Immunogenicity endpoints: anti-SHR-1819 antibody (ADA) positive rate and onset time. | 1-85 days

IPD SHARING:
Plan to Share IPD: Undecided